CLINICAL TRIAL: NCT06169800
Title: A Pilot Study to Evaluate the Effectiveness of a Biologic Augment of the Medial Patellofemoral Ligament to Reduce Recurrence After a Primary Lateral Patellofemoral Dislocation (BioPPD)
Brief Title: Biologic Augment of the Medial Patellofemoral Ligament Following Primary Lateral Patellofemoral Dislocation (BioPPD)
Acronym: BioPPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Banff Sport Medicine Foundation (Other)
Collaborators: CONMED Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB23-1095
Record Dates: First submitted 2023-12-05; First posted 2023-12-14 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-01

CONDITIONS: Patellofemoral Dislocation

STUDY DESIGN:
Intervention Model Description: This investigator-initiated pilot trial will assess patients with a first-time lateral patellofemoral dislocation following surgical MPFL repair augmented with a Biobrace®. Patients will be evaluated for two years post-operative, using patient-reported outcome measures and objective clinical and functional testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- MPFL repair with Biobrace augmentation (Experimental): Patients presenting with first-time lateral patellofemoral dislocation within the previous 7 days will be offered a patellofemoral stabilization procedure, including knee arthroscopy and an MPFL repair augmented with Biobrace® synthetic ligament.
  Interventions: Device: MPFL repair with Biobrace augmentation

INTERVENTIONS:
Device: MPFL repair with Biobrace augmentation — MPFL repair with Biobrace augmentation

SUMMARY:
This study aims to determine the ability of medial patellofemoral ligament (MPFL) repair augmented with Biobrace® to decrease the re-dislocation rate after a primary patellofemoral dislocation. First-time patellofemoral dislocation is a significant problem, and the ramifications of recurrence for patients are substantial. Due to the multifactorial nature of the pathoanatomy of patellofemoral instability, it has been difficult to design trials that will show how interventions could affect the natural history of these young patients. No definitive studies have determined whether the surgical reconstruction of the MPFL in patients with mild to moderate pathoanatomic risk factors will decrease the re-dislocation rate after a first-time dislocation. In addition, to date, no synthetic option has provided both biology and strength for ligament augmentation. This innovation may allow for a minimalist approach to keeping the patella centred in the trochlear groove during the healing phase after a first-time dislocation.

DETAILED DESCRIPTION:
This study aims to determine the ability of MPFL repair augmented with Biobrace® to decrease the re-dislocation rate after a primary patellofemoral dislocation. The null hypothesis is that there will be no difference in re-dislocation rate 2 years after surgical stabilization with Biobrace® compared to the natural history of patellar instability.

Patellofemoral instability is a well-recognized and common knee joint injury. Studies reporting the natural history after a first-time patellofemoral dislocation have reported a recurrence rate ranging from 10-80%. Recurrence varies depending on the unique pathoanatomic risk factors of each patient. Risk factors related to recurrence after a first-time dislocation include open growth plates, age at first dislocation, trochlear dysplasia, increased tibial tubercle - trochlear groove (TT-TG) distance, contralateral dislocation, and patella alta. A recent systematic review and meta-analysis determined the redislocation rate in patients managed without surgery after a first-time dislocation was 30%.

The MPFL plays a critical role in the constraint of lateral translation of the patella, providing 50-60% of the soft tissue restraint in early flexion before the patella engages in the trochlear groove. Essentially, the MPFL guides and holds the patella in the trochlear groove, especially between 0-45 degrees of flexion. MPFL insufficiency is present in as many as 90% of acute patellar dislocations and up to 100% of recurrent cases. The traditional non-operative treatment for a first-time dislocation has been to splint the knee in extension, which may prevent further dislocation but does not reduce the patella in the trochlear groove so that the medial soft tissue can heal in an anatomic position.

Multiple studies have investigated operative and non-operative treatments that aim to reduce recurrence after a first-time patellofemoral dislocation. To date, the type of knee immobilization has not been demonstrated to influence the recurrence rate. Operative management has been investigated compared to traditional non-operative treatment. A systematic review tabulated 15 studies comparing MPFL repair to non-operative management demonstrated decreased re-dislocation rates and decreased knee pain in those with surgical repair. Liebensteiner et al. reviewed studies with level 1 or 2 evidence and concluded that there are mixed results and that consensus on the ideal management after a first-time dislocation is still unclear. Despite these published results, surgical treatment after a first-time dislocation has not found widespread acceptance.

Further trials have compared MPFL repair to MPFL reconstruction. Bitar et al. conducted a study of MPFL reconstruction compared to non-operative management using the current a la carte indications for isolated MPFL reconstruction. These authors concluded that MPFL reconstruction was superior for preventing re-dislocation of the patella. Another recent retrospective review of 76 patients with an osteochondral lesion followed for 2 years compared MPFL-R to MPFL repair or no treatment. This study determined that completing an MPFL-R at index surgery resulted in a 5-fold reduction in recurrent instability.

Synthetic products can be used as a graft to reconstruct an MPFL. A systematic review has reported good results at a minimum of 2 years post-operative. Most synthetic products available today to augment or enhance the repair of ligaments are designed to address only one of two failure mechanisms: they either add mechanical strength without biological healing or aid in remodelling the underlying tendon tissue without providing mechanical strength during surgical repair. The inability of current devices to both strengthen the repair and create a favourable healing environment for cellular infiltration and tissue growth has led to further innovation and the development of the Biobrace® implant by Biorez. The Biobrace® implant is intended for use in general surgical procedures to reinforce soft tissue where weakness exists. The Biobrace® implant is also designed to reinforce soft tissues repaired by suture or suture anchors during tendon or ligament repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 - 30 years
* First-time lateral patellofemoral dislocation in the previous 7 days
* Closed or closing growth plates (confirmed on knee x-rays with no change required for surgical technique)

Exclusion Criteria:

* History of previous patellofemoral dislocation on the index knee
* An osteochondral fracture of the patellofemoral joint that requires surgical repair
* Unable to complete computer-based outcome questionnaires
* Pregnant at the time of surgery

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrent Dislocation of the Patella | 2-years
  Reports of patellar dislocation will be recorded during the follow-up visits, and a clinical assessment of patellar mobility will be completed to assess the integrity of the MPFL to confirm the redislocation. The rate of re-dislocation will be calculated and compared with the published 30% recurrence rate for patients managed conservatively following a first-time patellar dislocation. A relative risk and risk difference of re-dislocation will be calculated.

SECONDARY OUTCOMES:
Banff Patellofemoral Instability Instrument (BPII 2.0) | 2-years
  The BPII 2.0 is a valid and reliable, disease-specific quality-of-life score with five domains, including symptoms and physical complaints; work-related concerns; sport, recreation, and competition; lifestyle; and social and emotional. This patient-reported outcome will be assessed before surgery, and 6, 12, and 24 months after surgery. Score range 0-100, with higher score indicative of higher quality of life.
Single-leg Hop tests | 2-years
  The hop tests involve a comparative assessment of limb-to-limb function for a single hop for distance, a 6-metre timed hop, a triple hop for distance, and a triple cross-over hop at 6, 12, and 24 months after surgery.
Single-leg Balance test | 2-years
  Single-leg balance on a Bosu ball will be assessed for each limb to a maximum time of 30 seconds at 6, 12, and 24 months after surgery.
Isometric Muscle Strength | 2-years
  A crane gauge will be used to measure quadriceps and hamstrings strength in kilograms before surgery and 6, 12, and 24 months after surgery.
Recurrent Instability of the Patella (RIP) Score | 2-years
  The RIP score uses age, skeletal maturity, trochlear dysplasia, and TT-TG/PL ratio to predict recurrence. This score can categorize patients into low, intermediate, and high risk for re-dislocation.
Visual analogue scale (VAS) pain scores in the initial 14-days post-operative | 2-weeks
  A log book will be used to record VAS pain scores twice daily for the first 14 days post-operative. The score will be marked on a 100mm line where o represents no pain and 100 represents severe pain.
Medication use in the initial 14-days post-operative | 2-weeks
  A log book will be used to record medication use for the first 14 days post-operative. Patients will indicate the medications used and the dose consumed each day.
Tampa Kinesiophobia Scale (TSK-11) | 2-years
  Patient-reported outcome measure of kinesiophobia using the TSK-11 will completed pre-operatively and 6, 12, and 24 months post-operative. The minimum score is 11 and the maximum score is 44, with higher scores indicative of greater kinesiophobia.
ACL Return to Sport after Injury (ACL-RSI) | 2-years
  Patient-reported outcome measure for return to sport using the ACL-RSI will completed pre-operatively and 6, 12, and 24 months post-operative. The minimum score is 0 and the maximum score is 100. Higher scores indicate greater psychological preparation for return to sport.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A Hiemstra, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Banff Sport Medicine, Canmore, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No